CLINICAL TRIAL: NCT06420349
Title: Phase 1b Study of the Novel GCN2 Kinase Activator NXP800 in Patients With Advanced Cholangiocarcionoma
Brief Title: NXP800 for the Treatment of Patients With Advanced or Metastatic Cholangiocarcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: study sponsor phasing out drug supply
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC230406; NCI-2024-03613 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC230406 (Other: Mayo Clinic); 23-012778 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-05-08; First posted 2024-05-20 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Advanced Cholangiocarcinoma; Metastatic Cholangiocarcinoma; Refractory Cholangiocarcinoma; Stage III Hilar Cholangiocarcinoma AJCC v8; Stage III Intrahepatic Cholangiocarcinoma AJCC v8; Stage IV Hilar Cholangiocarcinoma AJCC v8; Stage IV Intrahepatic Cholangiocarcinoma AJCC v8
MeSH Terms: conditions — Cholangiocarcinoma; Klatskin Tumor | interventions — Specimen Handling; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (NXP800) (Experimental): Patients receive NXP800 according to assigned treatment schedule. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT, MRI, and/or PET at baseline and on study. Patients may optionally undergo ultrasound-guided tumor biopsy and/or collection of blood samples on study and during follow up.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Heat Shock Factor 1 Pathway Inhibitor NXP800; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Procedure: Ultrasound-Guided Biopsy

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Biological: Heat Shock Factor 1 Pathway Inhibitor NXP800 — Given PO
  Other Names: CCT 361814; CCT-361814; CCT361814; HSF1 Pathway Inhibitor NXP800; NXP-800; NXP800; VK2019
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Procedure: Ultrasound-Guided Biopsy — Undergo ultrasound-guided tumor biopsy
  Other Names: Ultrasound Biopsy; Ultrasound Guided Biopsy

SUMMARY:
This phase I trial tests the safety, best dose, and effectiveness of NXP800 in treating patients with cholangiocarcinoma that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced) or that has spread from where it first started (primary site) to other places in the body (metastatic). NXP800 inhibits a pathway called the heat shock factor 1 (HSF1) pathway. The inhibition of this pathway inhibits proliferation, migration, survival, and metastasis in susceptible tumor cells. Overexpressed, amplified and/or overactivated in many cancer cells, HSF1 activates a set of genes that play a key role in tumor initiation, progression and metastasis. Inhibiting this pathway may in turn inhibit tumor initiation, progression, and/or metastasis. Giving NXP800 may be safe, tolerable and/or effective in treating patients with advanced or metastatic cholangiocarcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the maximum tolerated dose (MTD)/recommended phase 2 dose for heat shock factor 1 pathway inhibitor NXP800 (NXP800).

SECONDARY OBJECTIVES:

I. To determine the toxicity profile of NXP800. II. To determine the best response for NXP800 using Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1.

III. To estimate the overall survival (OS) for NXP800. IV. To estimate the progression-free survival (PFS) for NXP800.

EXPLORATORY OBJECTIVES:

I. To evaluate transcriptomic features associated with sensitivity, resistance and pharmacodynamic effect of NXP800 using serial ribonucleic acid-sequencing (RNA-Seq).

II. To assess tumor evolution with NXP800 using serial whole genome-sequencing (Seq).

III. To assess tumor evolution with NXP800 using serial circulating tumor deoxyribonucleic acid (DNA) (ct-DNA).

IV. To estimate tumor marker response using serial CA19-9/carcinoembryonic antigen (CEA).

OUTLINE: This is a dose de-escalation study of NXP800 followed by a dose-expansion study.

Patients receive NXP800 orally (PO) according to assigned treatment schedule. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT), magnetic resonance imaging (MRI), and/or positron emission tomography (PET) at baseline and on study. Patients may optionally undergo ultrasound-guided tumor biopsy and/or collection of blood samples on study and during follow up.

After completion of study treatment, patients are followed up every 6 months until progressive disease or death for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically/cytologically confirmed biliary tract cancer
* Advanced or metastatic disease that is refractory to gemcitabine or fluoropyrimidine based therapy, or if there is intolerance to these regimens
* Measurable disease by RECIST 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Anticipated life expectancy of > 12 weeks
* Hemoglobin ≥ 9.0 g/dL (obtained ≤ 14 days prior to registration)
* Absolute neutrophil count (ANC) ≥ 1500/mm^3 (obtained ≤ 14 days prior to registration)
* Platelet count ≥ 100,000/mm^3 (obtained ≤ 14 days prior to registration)
* Aspartate aminotransferase (AST) ≤ 5 x upper limit of normal (ULN) (obtained ≤ 14 days prior to registration)
* Alanine aminotransferase (ALT) ≤ 5 x ULN (obtained ≤ 14 days prior to registration)
* Total bilirubin ≤ 1.5 x ULN (obtained ≤ 14 days prior to registration)
* Serum creatinine ≤ 1.5 x ULN (obtained ≤ 14 days prior to registration)
* Provide written informed consent
* Negative pregnancy test done ≤ 7 days prior to registration, for persons of childbearing potential only

  * NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Willing to use a highly effective method of contraception from the first dose of study medication through 180 days after the last dose of study medication, for persons of childbearing potential or persons able to father a child only
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)

Exclusion Criteria:

* Any of the following because this study involves an investigational agent whose genotoxic, mutagenic, and teratogenic effects on the developing fetus and newborn are unknown:

  * Pregnant persons.
  * Nursing persons.
  * Persons of childbearing potential who are unwilling to employ adequate contraception
* Systemic anti-neoplastic therapy or radiation therapy ≤ 14 days prior to registration
* Major surgical procedure ≤ 28 days prior to registration
* Ongoing therapy related events > grade 2
* Presence of another primary malignancy not in remission
* New York Heart Classification 3 or greater heart failure
* QT/corrected QT (QTc) interval > 470 ms using Fredericia's QT correction formula
* Uncontrolled brain metastatic disease
* Uncontrolled infection
* Any other comorbidities within the opinion of the investigator interfere with the investigation of the protocol
* Usage of drugs that strongly inhibit or induce CYP3A4 ≤ 7 days prior to registration and for the duration of NXP800 dosing. Drugs that are low, medium, or other inhibitors of CYP3A4 are not prohibited and should be used with caution. Drugs that inhibit BCRP are not prohibited but should be used with caution, since NXP800 was found to be a BCRP substrate
* Usage of seville oranges, grapefruit or grapefruit juice or products ≤ 7 days prior to registration and for the duration of NXP800 dosing
* Unwillingness to follow study related procedures
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2024-05-31 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 12 months
  MTD is defined as the dose level below the lowest dose that induces dose-limiting toxicity in at least one-third of patients.
Recommended phase 2 dose | Up to 12 months
  Recommended phase 2 dose is based on MTD (Outcome 1).

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 30 days after the administration of the last dose of study drug
  Overall toxicity incidence as well as toxicity profiles by dose level, patient and tumor site will be explored and summarized. Frequency distributions, graphical techniques and other descriptive measures will form the basis of these analyses. The grade 3+ adverse events will also be described and summarized in a similar fashion.
Best response | Up to 3 years
  Best response is defined to be the best objective status recorded. The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria. The Response Evaluation Criteria in Solid Tumors 1.1 criteria will be used for tumor evaluation and patients will be re-evaluated every 8 weeks. Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease in this patient population (overall and by dose level). The number of responses may indicate further evaluation for specific tumor types in a phase II setting.
Overall survival (OS) | Up to 3 years
  OS will be estimated using the Kaplan-Meier method. The median OS and corresponding 95% confidence interval (by Brookmeyer and Crowley) will be reported.
Progression-free survival (PFS) | Up to 3 years
  PFS will be estimated using the Kaplan-Meier method. The median PFS and corresponding 95% confidence interval (by Brookmeyer and Crowley) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh J. Borad, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- [Derived] Kuipers H, Larson JJ, Conboy CB, Ahn DH, Bekaii-Saab T, Wu C, Sonbol MB, Ilyas SI, Gores GJ, Smoot RL, Borad MJ. A Phase 1 study of the novel GCN2 kinase activator NXP800 in patients with advanced cholangiocarcinoma. Future Oncol. 2025 Sep;21(21):2723-2730. doi: 10.1080/14796694.2025.2539611. Epub 2025 Jul 28. PMID 40717483
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials